CLINICAL TRIAL: NCT01154179
Title: Appropriate Controlled Feeding: a Single Blinded Prospective Randomised Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scarborough General Hospital (Other)
Responsible Party: Principal Investigator, Anwar Owais, Mr, Scarborough General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SNE-A01322
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Patients Requiring Artificial Nutrition
Keywords: permissive underfeeding; hypocaloric feeding; artificial nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Normocaloric feeding (No Intervention): This control group will receive energy and protein intakes as recommended by the use of Schofield equations, as is current practice (100% of requirements)
  Interventions: Other: Hypocaloric feeding

INTERVENTIONS:
Other: Hypocaloric feeding — This intervention group will be prescribed 60% of recommended (by Schofield) requirements.

SUMMARY:
During patients' stay in the hospital, some of the patients may require artificial feeding for various reasons either through a vein or through a tube going directly to the gut. However, the amount of feeding that can be considered 'adequate' is unclear due to lack of research data. The current evidence the investigators have suggests that doctors might be giving patients more than they require, which might carry some risks. This hasn't been proven until now and there is no evidence as yet to show investigators exactly how much the doctors should feed patients.

The aim of the study is to see whether feeding patients less than what they are currently been feed is associated with better outcome.

The patients will be randomly (like tossing a coin) allocated into 2 groups. One group will get 100% of the current amount; the second group will get 60%. The investigators will then compare the groups to decide if feeding patients less than the current practice is associated with better outcomes.

DETAILED DESCRIPTION:
Aims:

The primary aim of this study is to assess whether hypocaloric feeding in patients receiving artificial nutritional support is associated with reduced septic and non septic morbidity compared to "standard" nutritional support. Secondary end points will include the assessment of metabolic, physiological and clinical responses to the different feeding protocols.

ENTERAL FEEDING OBJECTIVES

1. To investigate whether or not hypocaloric feeding in patients receiving enteral artificial nutritional support is associated with reduced septic and non septic morbidity compared to "standard" nutritional support.
2. To investigate whether or not hypocaloric feeding in patients receiving enteral artificial nutritional support is associated with changes in the inflammatory response compared to "standard" nutritional support.
3. To investigate whether or not hypocaloric feeding in patients receiving enteral artificial nutritional support is associated with changes in metabolic response compared to "standard" nutritional support.
4. To investigate whether or not hypocaloric feeding in patients receiving enteral artificial nutritional support is associated with changes in nutrition status compared to "standard" nutritional support.
5. To investigate whether or not hypocaloric feeding in patients receiving enteral artificial nutritional support is associated with differences in systemic complications compared to "standard" nutritional support.
6. To undertake a cost benefit analysis in patients receiving enteral artificial nutritional support, with the assumption that patients receiving hypocaloric feeding will not necessarily manifest lower feeding costs.

PARENTERAL FEEDING OBJECTIVES

1. To investigate whether or not hypocaloric feeding in patients receiving parenteral artificial nutritional support is associated with reduced septic and non septic morbidity compared to "standard" nutritional support.
2. To investigate whether or not hypocaloric feeding in patients receiving parenteral artificial nutritional support is associated with changes in the inflammatory response compared to "standard" nutritional support.
3. To investigate whether or not hypocaloric feeding in patients receiving parenteral artificial nutritional support is associated with changes in metabolic response compared to "standard" nutritional support.
4. To investigate whether or not hypocaloric feeding in patients receiving parenteral artificial nutritional support is associated with changes in nutrition status compared to "standard" nutritional support.
5. To investigate whether or not hypocaloric feeding in patients receiving parenteral artificial nutritional support is associated with differences in systemic complications compared to "standard" nutritional support.
6. To undertake a cost benefit analysis in patients receiving parenteral artificial nutritional support, with the assumption that patients receiving hypocaloric feeding will not necessarily manifest lower feeding costs.

Study Design and Study Group:

This will be a single blind, randomized controlled clinical trial. All patients requiring adjuvant nutritional support will be included in this study. The need for nutritional support and the method of administration (enteral or parenteral) will be decided by the hospital's nutrition team as is present practice.

Clinically, patients requiring supplemental nutrition fall into two clinical groups. Those with a functional gut are fed enterally; the other group, whose gut, for whatever reason, is not functional are fed parenterally. This is the rationale of studying two groups of administration.

Please see Flowchart for exact details. Patients will enter into the parenteral or the enteral component of the stud y in a mutually exclusive manner with no crossover or randomisation occurring at this point. Thereafter, patients in either arm of the study (enteral or parenteral) will be randomised to one of two groups. Comparisons will be done within, but not across, each of the enteral and parenteral arms.

Enteral feeding details:

Enteral control group: patients will receive energy and protein intakes as recommended by the use of Schofield equations (TER=total energy requirements), as is current practice.

Enteral intervention group: patients will be prescribed 60% of recommended (by Schofield) requirements.

Parenteral feeding details:

Parenteral control group : the control group, will receive energy and protein intakes as recommended by the use of Schofield equations, as is current practice.

Parenteral intervention group: patients will be prescribed 60% of recommended (by Schofield) requirements.

Data analysis will be on an "intention to treat" basis. Enteral and parenteral study arms will be analysed separately.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring artificial nutritional support in the hospital

Exclusion Criteria:

* Failure to obtain informed consent / assent from next of kin.
* Patients at risk of refeeding syndrome.
* If patients require concomitant enteral and parenteral nutrition.
* Pregnant women and children under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Septic complication | average of one week

SECONDARY OUTCOMES:
Inflammatory response | average of one week
Metabolic response | average of one week
Nutrition status | average of one week
Systematic complications | average of one week
Cost benefit analysis | average of one week

CONTACTS AND LOCATIONS:
Overall Officials: Anwar E Owais, MBBS MRCSEd, Principal Investigator — Scarborough General Hospital; Irfan Kabir, MRCS, Principal Investigator — SCarborough General hopital; Marcel Gatt, MD, Principal Investigator — Scarborough General Hospital; Claire Mcnaught, MD, Principal Investigator — Scarborough General Hospital; John Macfie, MD, Principal Investigator — Scarborough General Hospital
Locations (1):
- Scarborough General Hospital, Scarborough, North Yorkshire, United Kingdom

REFERENCES:
- [Derived] Owais AE, Kabir SI, Mcnaught C, Gatt M, MacFie J. A single-blinded randomised clinical trial of permissive underfeeding in patients requiring parenteral nutrition. Clin Nutr. 2014 Dec;33(6):997-1001. doi: 10.1016/j.clnu.2014.01.005. Epub 2014 Jan 12. PMID 24467878